CLINICAL TRIAL: NCT00798603
Title: A Phase II First-Line Study of a Combination of Pemetrexed, Carboplatin and Bevacizumab in Advanced Nonsquamous NSCLC Evaluating Efficacy and Tolerability in Elderly Patients (Age ≥ 70 Yrs) With Good Performance Status (PS < 2)
Brief Title: Pemetrexed, Carboplatin, and Bevacizumab as First-Line Therapy in Treating Older Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0821; NCI-2009-00670 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000626346 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Results first posted 2017-01-25 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Bevacizumab; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pemetrexed + carboplatin + bevacizumab (Experimental): Patients receive pemetrexed disodium IV over 10 minutes, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease or partial or complete response after 6 courses may continue to receive pemetrexed disodium and bevacizumab every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: pemetrexed disodium

INTERVENTIONS:
Biological: bevacizumab
Drug: carboplatin
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Pemetrexed may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving pemetrexed together with carboplatin and bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving pemetrexed together with carboplatin and bevacizumab works as first-line therapy in treating older patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the progression-free survival at 6 months in elderly patients with advanced nonsquamous cell non-small cell lung cancer treated with pemetrexed disodium, carboplatin, and bevacizumab as first-line therapy.

Secondary

* To assess the adverse events profile and safety of this regimen in these patients.
* To estimate the confirmed antitumor response rate, as defined by RECIST criteria, and the overall survival of these patients.
* To compare the quality of life (QOL) of patients treated with this regimen vs the QOL of younger patients.
* To correlate QOL with toxicities, as defined by NCI CTCAE v3.0 criteria.

Tertiary

* To evaluate polymorphisms in the genes that encode proteins involved in the cellular transport, activation, and cytotoxic activity of pemetrexed disodium and evaluate their relationship with treatment toxicity/efficacy and patient QOL.
* To evaluate polymorphisms in the genes involved in blood pressure regulation and their relationship with susceptibility to hypertension induced by anti-VEGF therapy.

OUTLINE: This is a multicenter study.

Patients receive pemetrexed disodium IV over 10 minutes, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable disease or partial or complete response after 6 courses may continue to receive pemetrexed disodium and bevacizumab every 21 days in the absence of disease progression or unacceptable toxicity.

Tissue and blood samples are collected at baseline for pharmacogenetic analysis. Blood samples are used to evaluate functionally relevant polymorphisms in the genes that encode proteins involved in the transport and activation of pemetrexed disodium and in the genes that encode proteins involved in susceptibility to hypertension induced by bevacizumab. Tissue samples are used to evaluate expression and polymorphisms in pemetrexed disodium target genes (TS, DHFR, and GARFT).

Quality of life is assessed at baseline and periodically during study.

After completion of study therapy, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed nonsquamous cell non-small cell lung cancer (NSCLC)

  * Stage IIIB (with pleural effusion) or IV disease
  * Squamous cell carcinomas not allowed

    * Adenosquamous histology allowed
* Clinically significant effusion (e.g., symptomatic pleural effusion or ascites) allowed provided it is drained before study treatment

  * No symptomatic pleural and/or peritoneal effusion (≥ grade 2 dyspnea, as defined by NCI CTCAE v3.0 criteria) that is not amenable to drainage
  * If effusion produces clinically significant measurable objective changes, such as hypoxia or estimated volume > 500 mL, effusion should be drained even if asymptomatic
* Measurable disease, defined as ≥ 1 lesion with longest diameter ≥ 2.0 cm by conventional techniques or ≥ 1.0 cm by spiral CT scan

  * If the sole site of disease is in a previously irradiated field, must have evidence of disease progression/recurrence within the irradiated field OR presence of a new lesion outside the irradiated field
* No symptomatic, untreated, or uncontrolled CNS metastases

  * CNS metastases that were previously treated with whole brain radiotherapy (WBRT) allowed
* Willing to enroll in NCCTG-N0392

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) OR direct bilirubin normal
* AST and ALT ≤ 3 times ULN (≤ 5 times ULN if liver has tumor involvement)
* Creatinine clearance ≥ 45 mL/min
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* Able to take folic acid, vitamin B_12 supplementation, or dexamethasone
* Able to complete questionnaire(s) alone or with assistance
* Willing to provide biologic specimens as required by the study
* Willing to return to NCCTG participating center for follow-up
* No clinically significant infection
* No serious, nonhealing wounds, ulcers, or bone fractures
* No seizure disorder
* No second primary malignancy within the past 5 years, except for any of the following:

  * Carcinoma in situ of the cervix
  * Nonmelanomatous skin cancer

    * History of melanoma allowed only if diagnosed and definitively treated ≥ 5 years ago with no subsequent evidence of recurrence
  * Low-grade (Gleason score ≤ 6) localized prostate cancer (no nodal involvement)
  * Previously treated stage I breast cancer
* No concurrent severe and/or uncontrolled medical condition, including any of the following:

  * Hypertension, labile hypertension, or history of poor compliance with antihypertensive medication
  * Angina pectoris
  * Congestive heart failure within the past 3 months, unless ejection fraction > 40%
  * Myocardial infarction within the past 6 months
  * Cardiac arrhythmia
  * Diabetes mellitus
  * Interstitial pneumonia or extensive, symptomatic interstitial fibrosis of the lung
  * Active or recent history of hemoptysis > ½ teaspoon per event
  * Ongoing or active infection
  * Psychiatric illness/social situation that would limit compliance with study requirements
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 12 months
* No diverticulitis within the past 12 months
* No stroke within the past 6 months
* No significant traumatic injury within the past 8 weeks
* Not at greater than normal risk of bleeding

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiotherapy to > 25% of bone marrow
* More than 2 weeks since prior radiotherapy and recovered (alopecia allowed)
* At least 2 weeks since prior WBRT
* At least 3 days since prior gamma knife radiosurgery (without WBRT) for brain metastases
* More than 4 weeks since prior administration of live or attenuated viral vaccine
* More than 8 weeks since prior major surgery (e.g., laparotomy) or open biopsy (> 4 weeks since minor surgery)

  * Insertion of a vascular access device allowed
* No prior chemotherapy or systemic therapy for advanced lung cancer, except neoadjuvant or adjuvant chemotherapy
* No NSAID's 2 days prior to (5 days for long-acting NSAID's), the day of, and 2 days following protocol treatment
* More than 12 months since prior neoadjuvant therapy, adjuvant therapy, systemic chemotherapy, chemoradiotherapy, immunotherapy, or biologic therapy
* No concurrent anticoagulants

  * Low-dose warfarin or heparin for deep venous thrombosis prophylaxis allowed

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-12; Primary Completion 2011-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace K. Dy, MD, Study Chair — Roswell Park Cancer Institute
Locations (217):
- United States (217):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-five (65) participants were enrolled between December 12, 2008 and October 1, 2010. Final analysis as of November 6, 2012, was reported.
Pre-assignment Details: Three participants who never received any study treatment are excluded from all analyses.
Groups:
- Pemetrexed + Carboplatin + Bevacizumab: Patients receive pemetrexed disodium IV over 10 minutes, carboplatin IV over 30 minutes, and bevacizumab IV over 30-90 minutes on day 1.
Period: Overall Study
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Started | 62
Completed | 27
Not Completed | 35
Not completed — Still on treatment as of 11/6/2012 | 1
Not completed — Withdrawal by Subject | 10
Not completed — Adverse Event | 22
Not completed — Physician Decision | 1
Not completed — Lack of insurance coverage | 1

BASELINE CHARACTERISTICS:
Population: All participants who received treatment.
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 62
Age, Continuous [Median (Full Range); unit: years] | 74.5 [70 to 86]
Gender [Count of Participants; unit: Participants]
  Female | 31
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 58
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 62
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 30
  1=Symptomatic and fully ambulatory | 32
Histologic type [Count of Participants; unit: Participants]
  Adenocarcinoma | 44
  Other | 18
Non-small-cell lung cancer stage (TNM 6th edition) [Count of Participants; unit: Participants] — Stage IIIB: The cancer is continuing to spread from the lungs to the lymph nodes or to nearby structures and organs, such as the heart, trachea and esophagus.
  Stage IV: The cancer has metastasized throughout the body and may now affect the liver, bones or brain.
  Participants
    Stage IIIB | 9
    Stage IV | 53

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 6 Months
Description: Estimated using the Binomial point estimator (number of successes divided by the total number of evaluable patients). A patient is classified as a success if alive and progression-free at 6 months.
Time Frame: 6 months
Population: The first 55 participants who met the eligibility criteria and have started the study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 55
percentage of participants | 60 [45.9 to 73]

2. Secondary Outcome: Proportion of Confirmed Tumor Response Defined as an Objective Status of Complete Response or Partial Response on Two Consecutive Evaluations
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  Complete Response (CR): disappearance of all target and non-target lesions and no new lesions.
  Partial Response (PR): disappearance of all target lesions, persistence of one or more non-target lesions, and no new lesions; or at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD, no appearance of one/more new lesions, unequivocal progression of existing non-target lesions, and no new lesions.
Time Frame: Duration of study until progression (up to 5 years)
Population: All participants who met the eligibility criteria, have started the study treatment and have post-baseline disease assessments.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 55
percentage of participants | 40 [27.0 to 54.1]

3. Secondary Outcome: Duration of Response
Description: Duration of response for responders was defined as the time from the date of the first objective status assessment of a confirmed CR or PR to the first date of disease progression. Duration of response will be censored at the date of last post-therapy follow-up visit for responders who have not had disease progression. Duration of response will be calculated for all evaluable patients who have achieved an objective confirmed response.
Time Frame: Up to 5 years
Population: All participants who met the eligibility criteria, have started the study treatment and had confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 22
months | 8.8 [3.8 to 20.9]

4. Secondary Outcome: Number of Grade 3 or Higher Adverse Events Occurring in >=10% of Patients
Description: Adverse events were assessed by Common Terminology Criteria for Adverse Events (CTCAE) v3.0. Grading: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening, Grade 5=Death.
Time Frame: Up to 2.5 years
Population: All participants who received treatment.
Measure: Number; unit: particpants
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 62
particpants
  Fatigue | 16
  Hypertension | 7
  Neutropenia | 18
  Thrombocytopenia | 11

5. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined to be the time from date of registration to the date at which the patient is removed from the treatment due to progression, toxicity, refusal or death from any cause.
Time Frame: Up to 5 years
Population: All participants who met the eligibility criteria and have started the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 57
months | 4.89 [3.88 to 6.37]

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from study enrollment to the first date of disease progression or death as a result of any cause, whichever occurs first. Progression-free survival will be censored at the date of the last contact for patients who are still alive and who have not had disease progression.
Time Frame: Up to 5 years
Population: All participants who met the eligibility criteria and have started the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 57
months | 7 [5.9 to 10.1]

7. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from study enrollment to the time of death from any cause. Overall survival will be censored at the date of the last follow-up visit for patients who are still alive or lost to follow-up.
Time Frame: Up to 5 years
Population: All participants who met the eligibility criteria and have started the study treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 57
months | 13.7 [9.4 to 16.8]

8. Secondary Outcome: Change From Baseline to Cycle 3 in Quality of Life (QOL) as Assessed by the Lung Cancer Symptom Scale
Description: Lung Cancer Symptom Scale (LCSS) consist of 9 items that assess the symptoms of lung cancer during the past days on a 10-points scale with 0 as no symptoms and 10 as worse symptoms. The individual item score was translated onto a 0-100 point scale with lower values indicating worse symptoms. An average of the aggregate score of all 9 items was used for a total score. Change from baseline to cycle 3 was calculated by subtracting the baseline scores from the scores at cycle 3.
Time Frame: Baseline and Cycle 3
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 3 LCSS data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 46
units on a scale | 1.1 [-25.6 to 25.6]

9. Secondary Outcome: Change From Baseline to Cycle 5 in Quality of Life (QOL) as Assessed by the Lung Cancer Symptom Scale
Description: Lung Cancer Symptom Scale (LCSS) consist of 9 items that assess the symptoms of lung cancer during the past days on a 10-points scale with 0 as no symptoms and 10 as worse symptoms. The individual item score was translated onto a 0-100 point scale with lower values indicating worse symptoms. An average of the aggregate score of all 9 items was used for a total score. Change from baseline to cycle 5 was calculated by subtracting the baseline scores from the scores at cycle 5.
Time Frame: Baseline and Cycle 5
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 5 LCSS data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 37
units on a scale | 1.1 [-21.1 to 33.3]

10. Secondary Outcome: Change From Baseline to Cycle 3 in Overall Quality of Life Assessed by Linear Analogue Self Assessment (LASA)
Description: The overall quality of life (QOL) question was on a 10-points scale with 0=as bad as it can be and 10=as good as it can be. The QOL scores was translated onto a 0 to 100 point scale, with lower values indicating worse symptoms. Change from baseline to cycle 3 was calculated by subtracting the baseline scores from the scores at cycle 3.
Time Frame: Baseline and Cycle 3
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 3 LASA data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 45
units on a scale | 0 [-50 to 100]

11. Secondary Outcome: Change From Baseline to Cycle 5 in Overall Quality of Life Assessed by Linear Analogue Self Assessment (LASA)
Description: The overall quality of life (QOL) question was on a 10-points scale with 0=as bad as it can be and 10=as good as it can be. The QOL scores was translated onto a 0 to 100 point scale, with lower values indicating worse symptoms. Change from baseline to cycle 5 was calculated by subtracting the baseline scores from the scores at cycle 5.
Time Frame: Baseline and Cycle 5
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 5 LASA data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 37
units on a scale | 0 [-60 to 100]

12. Secondary Outcome: Change From Baseline to Cycle 3 in Fatigue Assessed by Treatment-specific Adverse Events Scale
Description: The single-item fatigue question was on a 10-points scale with 0=no fatigue and 10=as bad as you can imagine. The item scores was translated onto a 0 to 100 point scale, with lower values indicating worse symptoms. Change from baseline to cycle 3 was calculated by subtracting the baseline scores from the scores at cycle 3.
Time Frame: Baseline and Cycle 3
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 3 fatigue data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 45
units on a scale | 0 [-50 to 50]

13. Secondary Outcome: Change From Baseline to Cycle 5 in Fatigue Assessed by Treatment-specific Adverse Events Scale
Description: The single-item fatigue question was on a 10-points scale with 0=no fatigue and 10=as bad as you can imagine. The item scores was translated onto a 0 to 100 point scale, with lower values indicating worse symptoms. Change from baseline to cycle 5 was calculated by subtracting the baseline scores from the scores at cycle 5.
Time Frame: Baseline and Cycle 5
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 5 fatigue data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 37
units on a scale | -10 [-60 to 40]

14. Secondary Outcome: Change From Baseline to Cycle 3 in Neuropathy Assessed by Treatment-specific Adverse Events Scale
Description: The single-item neuropathy question was on a 10-points scale with 0=no numbness or tingling in fingers and toes and 10=worst numbness or tingling in fingers and toes imaginable. The item scores was translated onto a 0 to 100 point scale, with lower values indicating worse symptoms. Change from baseline to cycle 3 was calculated by subtracting the baseline scores from the scores at cycle 3.
Time Frame: Baseline and Cycle 3
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 3 neuropathy data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 45
units on a scale | 0 [-50 to 60]

15. Secondary Outcome: Change From Baseline to Cycle 5 in Neuropathy Assessed by Treatment-specific Adverse Events Scale
Description: The single-item neuropathy question was on a 10-points scale with 0=no numbness or tingling in fingers and toes and 10=worst numbness or tingling in fingers and toes imaginable. The item scores was translated onto a 0 to 100 point scale, with lower values indicating worse symptoms. Change from baseline to cycle 5 was calculated by subtracting the baseline scores from the scores at cycle 5.
Time Frame: Baseline and Cycle 5
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 5 neuropathy data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 37
units on a scale | 0 [-60 to 50]

16. Secondary Outcome: Change From Baseline to Cycle 3 in Nausea Assessed by Treatment-specific Adverse Events Scale
Description: The single-item nausea question was on a 10-points scale with 0=no nausea and 10=as bad as you can imagine. The item scores was translated onto a 0 to 100 point scale, with lower values indicating worse symptoms. Change from baseline to cycle 3 was calculated by subtracting the baseline scores from the scores at cycle 3.
Time Frame: Baseline and Cycle 3
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 3 nausea data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 45
units on a scale | 0 [-70 to 40]

17. Secondary Outcome: Change From Baseline to Cycle 5 in Nausea Assessed by Treatment-specific Adverse Events Scale
Description: The single-item nausea question was on a 10-points scale with 0=no nausea and 10=as bad as you can imagine. The item scores was translated onto a 0 to 100 point scale, with lower values indicating worse symptoms. Change from baseline to cycle 5 was calculated by subtracting the baseline scores from the scores at cycle 5.
Time Frame: Baseline and Cycle 5
Population: All participants who met the eligibility criteria, have started the study treatment and had baseline and cycle 5 nausea data.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Number analyzed (Participants) | 37
units on a scale | 0 [-90 to 20]

ADVERSE EVENTS:
Time Frame: 2.5 years
Arm/Group | Pemetrexed + Carboplatin + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 10/62
Other Adverse Events (participants affected / at risk) | 62/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin + Bevacizumab (N=62)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin + Bevacizumab (N=62)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 19 (48)
Hemolysis (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (2)
Dry eye syndrome (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 17 (25)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (26)
Diarrhea (Gastrointestinal disorders) | 24 (113)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 19 (39)
Flatulence (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Jejunal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 22 (66)
Nausea (Gastrointestinal disorders) | 40 (108)
Rectal pain (Gastrointestinal disorders) | 1 (2)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (38)
Disease progression (General disorders) | 2 (2)
Edema limbs (General disorders) | 1 (2)
Fatigue (General disorders) | 60 (444)
Fever (General disorders) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 3 (4)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 12 (23)
Lymphocyte count decreased (Investigations) | 6 (28)
Neutrophil count decreased (Investigations) | 46 (148)
Platelet count decreased (Investigations) | 45 (172)
Weight loss (Investigations) | 7 (24)
Anorexia (Metabolism and nutrition disorders) | 11 (23)
Blood glucose increased (Metabolism and nutrition disorders) | 10 (16)
Dehydration (Metabolism and nutrition disorders) | 7 (9)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 23 (84)
Seizure (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 2 (7)
Protein urine positive (Renal and urinary disorders) | 19 (54)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (33)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 9 (29)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 27 (128)
Hypotension (Vascular disorders) | 3 (3)
Peripheral ischemia (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less